CLINICAL TRIAL: NCT02109783
Title: Genetic Modifiers of Caffeine Intake and Athletic Performance
Brief Title: Caffeine, Genetic Variation and Athletic Performance
Acronym: GMC-AP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Nutrigenomix Inc. (Industry)
Responsible Party: Principal Investigator, Ahmed El-Sohemy, Associate Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 4168733312-CAF
Record Dates: First submitted 2014-04-03; First posted 2014-04-10 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
Keywords: Athletes; Ergogenic aids; Caffeine; Nutrigenomics; Genotype
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Caffeine 4 mg (Active Comparator): To compare exercise performance of 2 or 4 mg of caffeine per kilogram of body weight to placebo within subjects. Subjects will perform 4 exercise tests.
  Interventions: Dietary Supplement: Caffeine 4 mg
- Caffeine 2 mg (Active Comparator): To compare exercise performance of 2 or 4 mg of caffeine per kilogram of body weight to placebo within subjects. Subjects will perform 4 exercise tests.
  Interventions: Dietary Supplement: Caffeine 2mg
- Caffeine 0 mg (Placebo Comparator): To compare exercise performance of 2 or 4 mg of caffeine per kilogram of body weight to placebo within subjects. Subjects will perform 4 exercise tests.
  Interventions: Dietary Supplement: Caffeine 0

INTERVENTIONS:
Dietary Supplement: Caffeine 2mg — Caffeine 2 mg versus 4 mg/kg or placebo
  Arms: Caffeine 2 mg
Dietary Supplement: Caffeine 4 mg — To compare exercise performance of 2 or 4 mg of caffeine per kilogram of body weight to placebo within subjects. Subjects will perform 4 exercise tests.
  Arms: Caffeine 4 mg
Dietary Supplement: Caffeine 0 — To compare exercise performance of 2 or 4 mg of caffeine per kilogram of body weight to placebo within subjects. Subjects will perform 4 exercise tests.
  Arms: Caffeine 0 mg

SUMMARY:
Numerous studies have investigated the effect of caffeine on athletic performance, but the findings have not been consistent. This is due, in part, to the differences in response that has been observed both within and between studies. Previous research in our lab has shown that genetic variations affecting caffeine metabolism modify the association between caffeine and heart disease. We hypothesize that the inconsistencies among studies relating caffeine and athletic performance may be due to genetic differences in caffeine metabolism or response. Male athletes will take part in an intervention of caffeine versus placebo, using a randomized double-blinded placebo-controlled design, which will test various exercise protocols (power, strength, anaerobic capacity, endurance) that are associated with performance across multiple sports. We will conduct a genome-wide association study, which is an approach that involves scanning for markers across the genomes of our study participants together, not individuals, to find genetic variations associated with a particular trait such as VO2 max, lactate clearance efficiency, muscle fiber type and changes in exercise performance following caffeine. We will also examine known genetic variations that are associated with caffeine metabolism and response, to determine if these genes also affect response to exercise after ingesting caffeine. Subjects will be paid $50.

DETAILED DESCRIPTION:
Research Methods and Design

Experimental Design:

This randomized, double-blinded, placebo controlled, within-subjects counter-measured study design will include 100 male athletes from a variety of sports. Females will not be included in this study because hormonal contraceptive use, which is common among female athletes, and the time of the menstrual cycle have a significant effect on caffeine metabolism and exercise test performance measures. Controlling for these factors would require a much larger pool of participants and require considerable resources and time. However, if the findings from the proposed research show promising results in men we would then aim to replicate those findings in female athletes.

Participants will complete 4 visits (~90-120 min each) in the Human Physiology Research Laboratory in the Goldring Center at the University of Toronto. All testing will take place Monday to Saturday at various times. Participants will be instructed to maintain their regular diet (pre-testing meals will be replicated for all visits) and sleeping habits, avoid strenuous activity 48 hours before each visit, and abstain from caffeine one week prior to the first visit and for the duration of the data collection (4 weeks).

Sample Size Calculation

Parameters:

Effect size = 0.25: Although a large effect size for the main treatment effect was found in previous research (0.38), it was decided that to be conservative, this trial would be powered to detect a small-medium effect size which is still of physiological importance. Additionally, we are interested in the effects between the two doses of caffeine which are assumed to be smaller than the main treatment effect. Therefore, a small-medium effect size was needed to ensure sufficient statistical power to make between-caffeine-effect conclusions for the time trial analysis. Finally, other parameters of assessment such as the Vertical Jump for power will likely have a smaller effects size than the time-trial as reported by Tucker et al. (2013) in a study on vertical jump performance in male basketball players. Therefore, a smaller effect size would be required to adequately power the study for all outcome measures (i.e. power, strength anaerobic, aerobic etc.)

* Alpha (error probability) = 0.025: In general, an alpha = 0.05 is the standard value to use for this parameter. However, in our study the participants will be enrolled in a number of independent trials, and therefore it was decided to use a lower alpha so as to take into account error that can arise from multiple comparisons such as by sport (power or endurance) plus genotype (risk or common variant).
* Power (1-Beta probability) = 0.8: The conventional value of 0.8 was used for power.
* Number of groups = 2: Number of stratifications required for genotype subgroup analysis
* Number of measurements = 4: The laboratory exercise tests
* Correlation among repeat measures = 0: Zero correlation between measurements was assumed.
* Sample Size = 74: Based on calculations 74 participants are required. We will recruit 100 athletes in order to account for possible withdrawal of up to 25%, without potentially compromising the statistical significance of our results. In addition, if we choose to use multiple comparisons (genotype + sport) we would benefit from a larger sample to minimize the drop in effect size.

Recruitment

Recruitment will be carried out at the University of Toronto, Ryerson and York University campuses, the Canadian Sport Institute of Ontario, and at local running/triathlon clubs by flyers posted in appropriate locations. A standardized email with study and contact information will also be sent to head coaches and/or program directors of sports teams/clubs (at all locations listed above) with eligible athletes, who can then choose to make their athletes aware of the study.

Parameters of Assessment

Physiological data collected by two trained kinesiologists, a PhD level exercise physiologist, one student assistant and Nanci Guest, the graduate student.

Anthropometric and Clinical Characteristics

* Resting systolic (SBP) and diastolic (DBP) blood pressure measurements, as well as pulse rate, will be taken twice, one minute apart. The mean of the two consecutive readings will be taken.
* Heart rate will be measured before all tests to ensure participant calmness and similar physiological state for all tests and test days.
* Heart rate will be monitored throughout the duration of the trials (Visit 2-4) by Polar Heart Rate Monitors (Polar Electro, Finland)
* Height will be measured to the nearest 0.1 cm using a wall-mounted stadiometer and body weight will be measured to the nearest 0.1 kg using a digital scale with participant wearing light clothing and without shoes.
* Body weight value will be used to determine 2 and 4 mg per kilogram of body mass dosages for caffeine treatments (plus a placebo dose) that will be ingested in random order (derived by research assistant and blinded to all investigators) during visits 2, 3 and 4, over the following three weeks.
* Body Composition will be assessed by a bioimpedence scale (BC-558 Ironman Segmental Body Composition Monitor)

Exercise Tests

Descriptive Characteristics

Maximal Aerobic Capacity will be assessed by a VO2 max test on a cycle ergometer. This test is part of descriptive data and will be used to determine resistance set in the time trial test (65% peak power). Participants will undergo a graded exercise test on a Monark cycle ergometer (Groningen, The Netherlands) until volitional fatigue. To determine maximal oxygen consumption (VO2Max), air samples will be analyzed for oxygen and carbon dioxide concentrations via an indirect open circuit spirometry system (Parvomedics, Metabolic Cart, Sandy, Utah). Subjects will be set up with a Polar Heart Rate monitor.

Four main outcome measures (power, strength, anaerobic and aerobic capacity)

* Muscular Power will be assessed using the Vertical Jump Test (VJT) as described previously (5). Participants will complete two attempts at each of two vertical jump tests on a force plate (AMTI,Watertown, MA, USA).

  1. squat jump (SJ): from a squatting position (knee angle: 90° approximately) in which no preliminary counter movement is performed;
  2. counter-movement jump (CMJ): from an upright standing position with a preliminary counter movement; There will be a 30 second rest period between jumps and the best score of two will be recorded.
* Strength (upper body) will be assessed using a Handgrip Dynamometer (Lafayette Instrument Company model 78010). The highest score after 3 trials will be recorded (in kg).
* Anaerobic Capacity will be assessed using the Wingate Anaerobic Test on a cycle ergometer (Ergomedic 849E, Monark, Sweden). Participants will cycle against a fixed resistance of 0.085kg / kg body mass. Three main measures will be recorded during the test:

  * Peak power (PP): a measure of maximal anaerobic power, or the maximum power output reached for a 5-second period during the first 10 seconds of the test. PP will be recorded in Watts (W) and W/kg.
  * Mean power (MP): a measure of anaerobic capacity, or the mean power output achieved during the 30-second test. MP will be recorded in W and W/kg.
  * Fatigue Index (FI): a measure of the rate of power decrease, or the difference between the highest 5-second power output and the lowest 5-second power output, divided by elapsed time. FI will be recorded as a percentage.
* Endurance/Aerobic Capacity and power output will be assessed by a Cycling Time Trial (TT). Participants will be instructed to complete a 10 km TT, carried out on a cycle ergometer (Monarch Sports and Medical, Vansbro, Sweden), as quickly as possible with no temporal, verbal, of physiological feedback.Time required to complete the test and average power output will be recorded on completion of each test.

Additional Tests during Exercise Testing

* Blood Lactate Testing. Immediately after the Wingate test participants will have their finger pricked with a disposable lancet to puncture the skin and obtain a capillary blood sample for analysis with the Lactate Pro analyzer (LT-1710, Arkray Inc, Kyoto, Japan)
* Rating of Perceived Exertion (RPE) - The Borg scale for RPE will be used to assess subjects' perception of fatigue.

Genotyping

Saliva samples will be collected during Visit 1 of exercise testing using the Oragene-500 kit for DNA isolation using standard procedures as described previously.We will conduct a genome-wide association study, which is an approach that involves scanning for markers across the genomes of our study participants together, not individuals, to find genetic variations associated with a particular trait such as VO2 max, lactate clearance efficiency, muscle fiber type and changes in exercise performance following caffeine. We will also examine known genetic variations that are associated with caffeine metabolism and response, to determine if these genes also affect response to exercise after subjects ingest caffeine.

Dietary Intake Assessment

Subjects will complete a 196-item semi-quantitative food frequency questionnaire to determine habitual caffeine intake as well as other dietary factors. Dietary intake information will be used to identify potential effect modifiers such as usual caffeine consumption.

Health, Lifestyle and Physical Activity Assessment

The General health, lifestyle and physical activity questionnaire (GHLPA) will include detailed questions on caffeine (e.g. intake habits, withdrawal effects etc), previously used in our lab, combined with a validated habitual physical activity/sport history questionnaire previously used to assess sport/physical activity in athletes.

Statistical Analysis

Analyses will be carried out using SAS (Version 9.2, NC, USA, 2009) statistical software. Briefly, we will report descriptive data (height, weight, age, blood pressure, caffeine intake and habits, body fat %, VO2max, years in sport, training hours per week, dietary assessment data and other lifestyle measures) comparisons between genotype groups using independent t-tests. Potential differences in VO2max, 10 km time trial, anaerobic capacity, lactate threshold, power and strength and rate of perceived exertion will be assessed using repeated measures analysis of variance (RMANOVA) with treatment as a within participants factor and genotype as a between-participants factor. For all RMANOVA procedures, posthoc tests will be performed using independent and dependent t-tests with a Bonferroni correction such that P< 0.05 will be required as the threshold for significance.

Experimental Procedure

Initial Screening - phone call or in-person visit

Potential participants will verify their sports participation and ability to commit to four 2-hour visits to the lab 7 days apart. Participants will be reminded of the importance of maintaining their regular diet. The importance of the required caffeine abstinence, including any caffeine-containing supplements for 7 days prior to the first visit and the duration of the study (4 weeks) will be emphasized and reiterated.

Visit 1 (~90 min)

The first visit to the laboratory will involve familiarization, and obtaining written informed consent from all participants after an explanation about the aims, benefits, and risks involved with the study. Participants will be informed that they are free to withdraw from the study at any time.

Each subject will complete an "exercise readiness" questionnaire (PAR-Q; Physical Activity Readiness Questionnaire) have descriptive and anthropometric data collected, including date of birth, height, body mass, and blood pressure, and they will also provide a saliva sample for DNA isolation and genotyping. During this first visit, maximal oxygen uptake (VO2 max; described below) will also be measured for descriptive baseline data, and to derive workload levels for experimental time trials on subsequent testing visits.

Visit 2, 3 and 4 (~120 min)

All three visits will be identical with the exception of the 20 min waiting period (then 10 min pre-testing warm-up begins) for serum concentration of caffeine levels to reach peak levels, where the participant will complete a different questionnaire or sit quietly with their own activity.

Upon arrival participants will have been randomly assigned (to maintain blinding) to ingest either the supplement at 2 or 4 mg of caffeine per kg body weight, or dextrose placebo (PLAC). Each participant will ingest the same number of capsules with identical color and size during each visit, whether it is 0, 2 or 4 mg/kg, in order to maintain double-blinding of treatment. Each subject will complete a questionnaire or sit quietly (e.g. reading, using e-devices etc.) while waiting for the first exercise test.

Exercise test protocol will be identical for visits 2, 3 and 4. After 20 min, participants will warm-up for 10 min and then carry out 4 exercise tests (commencing at 30 min post-caffeine ingestion) to determine different measures of performance:

i. Muscle power - Vertical Jump Test

ii. Strength - Handgrip Dynamometer

iii. Anaerobic Capacity - Wingate

iv. Endurance/Aerobic Capacity (aerobic power) - 10 km Cycling Time Trial

Participants may drink water ad libitum throughout the exercise tests.

ELIGIBILITY:
Inclusion Criteria:

* healthy 18-35 yrs
* athlete competing/training in given sport 3 or more years
* currently competing at Varsity, Professional, National level or recreationally but also competing

Exclusion Criteria:

* medical conditions affected by caffeine / avoidance of caffeine
* injured / not training
* unable to abstain from caffeine for 4 weeks during study

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of caffeine to improve power, strength and speed | 2 hours
  To determine if their is a positive effect (improvement) effect of 2 or 4 mg of caffeine per kilogram of body mass on four distinct components of fitness: power, strength, anaerobic and aerobic capacity. Therefore, to determine the efficacy of caffeine to shorten time to completion in time trial, and increase power/strength in wingate, vertical jump and handgrip tests.

SECONDARY OUTCOMES:
Individual genotypes, caffeine ingestion and athletic performance | 1 day
  Saliva samples will be taken for a genome-wide association scan (GWAS) and identification of genetic variations related to caffeine metabolism, in order to determine which genes are associated with improved performance during the caffeine treatment. Sport SNP's on genes such as ACE, ACTN3 and others will also be identified to determine associations to performance and/or descriptive statistics such as VO2 max.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed El-Sohemy, PhD, Principal Investigator — University of Toronto
Locations (1):
- University ofToronto, Toronto, Ontario, Canada

REFERENCES:
- [Background] Tucker MA, Hargreaves JM, Clarke JC, Dale DL, Blackwell GJ. The effect of caffeine on maximal oxygen uptake and vertical jump performance in male basketball players. J Strength Cond Res. 2013 Feb;27(2):382-7. doi: 10.1519/JSC.0b013e31825922aa. PMID 22561972
- [Derived] Sicova M, Guest NS, Tyrrell PN, El-Sohemy A. Caffeine, genetic variation and anaerobic performance in male athletes: a randomized controlled trial. Eur J Appl Physiol. 2021 Dec;121(12):3499-3513. doi: 10.1007/s00421-021-04799-x. Epub 2021 Sep 16. PMID 34529114
- [Derived] Thakkar D, Sicova M, Guest NS, Garcia-Bailo B, El-Sohemy A. HFE Genotype and Endurance Performance in Competitive Male Athletes. Med Sci Sports Exerc. 2021 Jul 1;53(7):1385-1390. doi: 10.1249/MSS.0000000000002595. PMID 33433155
- [Derived] Guest NS, Corey P, Tyrrell PN, El-Sohemy A. Effect of Caffeine on Endurance Performance in Athletes May Depend on HTR2A and CYP1A2 Genotypes. J Strength Cond Res. 2022 Sep 1;36(9):2486-2492. doi: 10.1519/JSC.0000000000003665. Epub 2020 Jun 17. PMID 32569126